ARM A – adult patient

# University of Minnesota Department of Pediatrics

#### CONSENT TO PARTICIPATE IN RESEARCH

# Study of Epidermal Grafting Using the CelluTome® Epidermal Harvesting System for the Treatment of Individual Lesions in Persons with Epidermolysis Bullosa (EB)

#### Principal Investigator:

Christen Ebens, MD, MPH

You are invited to participate in this study because you had a stem cell transplant for Epidermolysis Bullosa (EB) which was successful but you still have areas of blistering skin that have not healed. This study is testing a method to heal these remaining areas of skin breakdown.

Taking part in any clinical research involves risks and may provide some benefits. You need to understand these risks and benefits to make an informed decision about whether or not to be in this study.

This form is called a consent form. The intent of this form is to let you know the purpose of this study and the possible risks and benefits of participation. If you wish to take part in this study, you will be asked to sign this consent form.

Research studies only include people who want to take part. Please take time to make your decision. We encourage you to discuss your decision with your doctors, family, and friends.

This study is being conducted at the University of Minnesota. Christen Ebens, MD, MPH in the Department of Pediatrics is the principal investigator (physician in charge) of this study.

August 10, 2021 HSC# 1512M81884 

ARM A - adult patient

#### Introduction

Areas of blistering (wounds) often remain even after a successful transplant. This study treats such areas by using covering the blistered area with a square of surgical tape (similar to 3M's Tegaderm® transparent dressing) that has been loaded with skin cells collected from the same donor as your transplant. The surgical tape is left on for 3-4 weeks to give the donor skin cells a chance to take hold and promote wound healing. It is like doing a skin graft, but only taking the top most layer of skin cells (the epidermis). The process is done in the out-patient clinic and is non-invasive and bloodless for both the person donating the skin cells and for the person receiving them. A summary of the donor collection process is attached at the end of this consent form.

The device used to collect the donor cells is the CelluTome Epidermal Harvesting System manufactured by KCI (an Acelity company). It was approved by the Food and Drug Administration in 2013 and is used for the treatment of chronic wounds including diabetic ulcers and bed sores. This study is unique in that it uses the donor from your original transplant to provide healthy skin cells. This is possible because donor cells from your original transplant are still present in your body as measured by blood and bone marrow chimerism (genetic profiles).

# Study Purpose

The primary goal of this study is to have partial to complete wound healing by 3 months after the epidermal cell graft in each of the treated areas. Secondary goals of the study include the appearance and health of the grafted skin 1 year later and to measure changes in quality of life (QOL) through a questionnaire created specifically for EB called iscorEB.

It is expected up to 60 people will be enrolled in this study with 40 of them using the donor from their previous transplant as the source of the skin cells (Arm A). The other 20 will have a patch of healthy skin as the source of the skin cells (Arm B) and will serve as their own donor.

# **Study Procedures**

To be considered for this study you must be at least 6 months out from transplant and meet all eligibility criteria as stated in the study. The person who served as your transplant donor must also be available and willing to provide skin cells. The donor (or

MT2015-36: Treatment of individual lesions in EB patients

ARM A - adult patient

parent/guardian if younger than 18 years) will be presented with a separate consent form which will be reviewed and written consent obtained if she/he agrees to be the skin cell donor for this study.

If you and the donor are eligible and agree to take part in this study, the following will occur.

You will have a brief physical exam (standard of care) and up to 3 areas of blistering will be identified for treatment (grafting) and an equal number areas will be identified but not treated at this time. The untreated areas are considered "controls." Photographs will be taken of each identified area.

The skin cells will be collected (harvested) from your donor according to the process summarized at the end of this consent. A different collection site will be used for each wound to be treated. Each harvest from the donor takes 30 to 40 minutes. At the end of each collection period, the harvested cells will be transferred onto a surgical tape patch.

The surgical tape then will be placed on one of the areas of blistering that were selected to be treated. Up to 3 donor skin cell transfers will be done during one clinic appointment with a separate surgical tape used for each. The surgical tape will be kept in place for 3 to 4 weeks to permit healing of heathy skin.

Photographs of each of the identified blistering areas will be taken once a week until your first follow-up appointment 6 weeks later. The photos will be done either in clinic or at home using a digital camera (such as a cell phone, iPad or camera) with the images sent to the University of Minnesota electronically by email or other photo sharing method.

Six weeks after the skin cell graft you and the donor may return to the University of Minnesota/or have a remote visit via phone call to have the collection sites (donor) and treated/control wounds (you) examined for healing. You will be asked to complete some brief questionnaires regarding your quality of life including pain and itch levels at each visit, also for research. Then, 12 weeks after the skin cell graft, you and the donor will return to the University of Minnesota/or have a remote visit via phone call to have the collection sites (donor) and treated/control wounds (you) examined for healing. You will be asked to complete another brief questionnaire regarding your quality of life including pain and itch, also for research. A final study visit occurs 1 year after the skin cell graft

MT2015-36: Treatment of individual lesions in EB patients

ARM A - adult patient

to see how well the treated areas have held up. This will include a physical exam and photographs of the sites.

While you are on this study you will also continue your previously planned post-transplant follow-up. Visits for both studies will be overlapped so you are not making separate visits for each study.

#### **Opportunity for Treatment of Additional Areas of Blistering:**

If at the 12 week (3 month) follow-up visit, the blister areas are healing well and your donor is willing, you may be offered treatment of the "control" wounds and/or other areas of blistering. This is optional and does allow for additional information to be collected for the study. You may have up to 3 sessions total with up to 3 blistering treated each time (9 wounds total). A new session must be at least 3 months from the previous session. As with the 1st treatment you will need to provide weekly photographs, but the 6 and 12 weeks clinic visits may be arranged at a medical facility closer to your home/or by a remote visit via phone call with the results sent to the University.

#### **Optional Skin Biopsy**

If you agree, we would like to take 3 additional samples of your skin, at a time when you are having a biopsy completed for clinical care purposes. These would be used for research tests that help determine whether the donor cells have "taken." Additionally, we would like to save any leftover cells for future research on EB. At the end of this document, you may opt in or opt out of having these samples collected and saved.

# **Length of Study Participation**

For the purpose of the study's research component, participation ends 1 year after the first treatment; however if you have additional skin collection sessions, information will continue to be collected until 1 year after the last session.

# **Risks of Study Participation**

There is a small amount of risk from participation in this study. If the donor cells do not take (non-engraftment) the cells will slough off because of low grade infection, inadequate blood supply or ongoing EB related fibrosis. If this occurs it may be accompanied by local inflammation and possibly fever (sign of a whole body reaction), although neither are expected to be serious.

August 10, 2021 HSC# 1512M81884 

ARM A - adult patient

In theory there is a risk of non-engraftment because the skin cells are being collected from a different person; however, since the skin cells come from the same donor as your transplant, you are essentially using your own cells since you share your donor's immune system.

The completion of the **iscorEB questionnaire** may remind you of the unpleasant aspects of your diagnosis. You may refuse to answer any questions that make you uncomfortable.

#### Risks associated with a skin biopsy:

Skin biopsy may cause pain, bleeding or bruising at the spot where the skin is taken. There may also be a small scar. Rare side effects include infection at the biopsy site, allergic reactions to the numbing medicine, and excessive scarring.

## **Benefits of Study Participation**

The intent is to provide long term healing of persistent areas of blistering although this is not known and the reason this study is being done. It is hoped that the findings in this study will improve the management of chronic areas of blistering for EB patients.

# **Alternatives to Study Participation**

You may choose to not participate in this study and continue with your current skin management plan.

# **Study Costs**

You are responsible for the costs of the procedures on this study, including the cost of the donor skin cell collection, the transfer of the donor cells to your areas of blistering, tests and physical examinations before and over the 1 year follow-up. Your insurance provider may not cover all or part of these costs. Preauthorization will be requested by a patient financial representative who will work with you and your nurse coordinator should your insurance company deny coverage. You should work with your patient financial representative as reimbursement – methods such as 3<sup>rd</sup> party reimbursement, charitable funds, self pay - must be confirmed prior to enrollment on this study. You will be responsible for any deductibles or co-pays.

You will receive no payment or compensation for taking part in this study.

August 10, 2021 HSC# 1512M81884 

ARM A – adult patient

#### **Research Related Injury**

In the event that this research activity results in an injury, treatment will be available, including first aid, emergency treatment and follow-up care as needed. Care for such injuries will be billed in the ordinary manner, to you or your insurance company.

It is important that you tell your study doctor or another member of the study staff if you feel that you have been injured because of taking part in this study. Dr. Ebens may be reached at 612-626-2961.

## Confidentiality

The records of this study will be kept private. Information will be kept in your electronic medical record, paper research chart and in study case report forms. Information gained from this study will be used for research and educational purposes. If information from this study is published or presented at scientific meetings, your name and other personal information will not be used.

Organizations that may look at and/or copy your medical records for research, quality assurance, and data analysis include:

- Departments at the University of Minnesota with appropriate regulatory oversight
- The Food and Drug Administration (FDA) and other governmental agencies involved in keeping research safe for people

To this extent, confidentiality is not absolute.

If you decide to participate in this study, some private health information about you will be stored in a computer database at the Masonic Cancer Center within the University of Minnesota. EB is not a cancer, but this database also stores information for non-cancer bone marrow transplants. This information will include your name and medical record number, date of birth, diagnosis, race/ethnicity, and information about your participation in this study. The purpose of storing this information is to assist the Cancer Center in creating reports about research and in making sure that research studies are being done correctly. Your information will not be used for any other purpose. There are no plans to erase information from the database. It will be stored indefinitely at the Masonic Cancer Center at the University of Minnesota.

August 10, 2021 HSC# 1512M81884 

MT2015-36: Treatment of individual lesions in EB patients

ARM A – adult patient

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. law. This website will not include information that could identify you. At most, the website will include a summary of the results. You may search this website at any time.

# **Protected Health Information (PHI)**

Your PHI created or received for the purposes of this study is protected under the federal regulation known as HIPAA. Refer to the attached HIPAA authorization for details concerning the use of this information.

## **Voluntary Participation**

Taking part in this study is your choice. You may choose either to take part or not to take part in the study.

If you decide to take part in this study, you may withdraw your consent at any time by contacting a member of the research staff. Any information obtained up to the time of withdrawal will continue to be used in the study's analysis.

No matter what decision you make, there will be no penalty to you and you will not lose any of your regular benefits. Leaving the study will not affect your medical care. You still may receive medical care from this institution.

## **New Information**

You will be told about new information or changes in the study that may affect your health or your willingness to continue in the study.

# **Contacts and Questions**

The physicians involved in your care are available to answer any questions you may have concerning this study at any time. Please ask any questions you have; we want you to understand the treatment and the study. If you have additional questions later concerning this study you are encouraged to call the study's Principal Investigator (lead physician) Dr. Christen Ebens at 612-626-2961.

August 10, 2021 HSC# 1512M81884 

ARM A – adult patient

Whom do I contact if I have questions, concerns or feedback about my experience? This research has been reviewed and approved by an IRB within the Human Research Protections Program (HRPP). To share feedback privately with the HRPP about your research experience, call the Research Participants' Advocate Line at 612-625-1650 (Toll Free: 1-888-224-8636) or go to z.umn.edu/participants.. You are encouraged to contact the HRPP if:

- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You want to talk to someone besides the research team.
- You have questions about your rights as a research participant.
- You want to get information or provide input about this research.

#### Will I have a chance to provide feedback after the study is over?

The HRPP may ask you to complete a survey that asks about your experience as a research participant. You do not have to complete the survey if you do not want to. If you do choose to complete the survey, your responses will be anonymous.

If you are not asked to complete a survey, but you would like to share feedback, please contact the study team or the HRPP. See the "Investigator Contact Information" of this form for study team contact information and "Whom do I contact if I have questions, concerns or feedback about my experience?" of this form for HRPP contact information.

August 10, 2021 HSC# 1512M81884 

| MT2015-36: | Treatment | of individual | lesions | in EB | patients |
|------------|-----------|---------------|---------|-------|----------|
|------------|-----------|---------------|---------|-------|----------|

ARM A – adult patient

# **Signature**

| l agree | l disagree | | | |
|---|---|---|---|---|
| | | The research may take two additional biopsies in order to determine who | | |
| | | With your permission, specimens have been completed may be sto that have not yet been determined be stored at the University of Minimused to develop new assay method in the event the samples are used they will be relabeled in an and identified in any way. The scientification the research to be done is not know will be informed of your individing treatment in any way. Some of the discoveries that may be of potentiand licensed for the development retain any property rights to the many money or other benefits that a or discoveries. Your decision not specimens will not affect your ability been read to me. I have had many you will be provided a copy of | red and used for future resid. Samples collected during nesota indefinitely. These sods for testing samples from d for tests outside the scopenymous manner, so that c, diagnostic and/or medicawn. Therefore, neither you rual results, and they will is research may result in neial commercial value and mit of new products. Donors aterials. Therefore, you wo may entity might receive for the allow storage or future us ity to participate in this study of questions answered. It a | earch purposes of the study may camples may be other subjects. See of this study, you cannot be a significance of nor your doctors not affect your ew inventions or may be patented of skin do not uld not share in these inventions see of your tissue you. |
| | | Signature Block for Capable | e Adult: | |
| | ature docume<br>is signed docu | nts your permission to take part in t | | ovided a |
| Signature | of Participant | | Date | |
| Printed N | ame of Particip | pant | | |
| Signature | of Person Ob | taining Consent | Date | |
| Printed N | ame of Persor | n Obtaining Consent | | |
| A 40 | 0004 | D0 | | |

August 10, 2021 HSC# 1512M81884 

Approved for use by UMN IRB Effective on 9/24/2021 IRB Study Number: 1512M81884

| MT2015-36: Treatment of individual lesions in EB patients | ARM A – adult patient |
|---|---|
| Signature Block for Witness: WITNESS STATEMENT: | |
| The participant was unable to read or sign this consen | t form because of the following reason: |
| ☐ The participant is unable to read the information | |
| ☐ The participant is visually impaired | |
| ☐ The participant is non-English speaking | |
| ☐ The participant is physically unable to sign the cons | ent form. Please describe: |
| ☐ Other (please specify): | |
| For the Consent of Non-English Speaking Participa As someone who understands both English and the la represent that the English version of the consent form subject's own language, and that the subject was given | nguage spoken by the subject, I was presented orally to the subject in the |
| Signature of Interpreter | Date |
| Printed Name of Interpreter OR: | |
| Statement from a Non-Interpreter: As someone who understands both English and the la that the English version of the consent form was prese own language, and that the subject was given the opportunity. | ented orally to the subject in the subject's |
| Signature of Individual | Date |
| Printed Name of Individual | |
| Signature Block for Adult Ur | nable to Consent: |
| Your signature documents your permission for the nan research. | ned participant to take part in this |
| Printed Name of Participant | |
| Average 40, 2024 | |

August 10, 2021 HSC# 1512M81884


| MT2015-36: Treatment of individual lesions in EB patients | ARM A – adult patient |
|---|---|
| Signature of Legally Authorized Representative | Date |
| Printed Name of Legally Authorized Representative Date | |
| Signature of Person Obtaining Consent | Date |
| Printed Name of Person Obtaining Consent Date | |

ARM A – adult patient



ARM A – adult patient

